CLINICAL TRIAL: NCT04361006
Title: Safety and Efficacy of Cryotherapy Versus Radiofrequency Ablation for Treatment of Para-hisian Accessory Pathways: a Randomized Comparative Trial
Brief Title: Cryotherapy Versus Radiofrequency Ablation for Treatment of Para-hisian Accessory Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Mauricio Ibrahim Scanavacca, Arrhythmia Unit Director - Heart Institute (InCor), MD, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4446/16/112; U1111-1250-5793 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Arrhythmias; Accessory Pathway; Wolf Parkinson White Syndrome
Keywords: para-hisian; radiofrequency; cryoablation; accessory pathway; electrophysiology
MeSH Terms: conditions — Arrhythmias, Cardiac; Pre-Excitation Syndromes; Wolff-Parkinson-White Syndrome | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Radiofrequency (RF) (Active Comparator): Twenty patients will be allocated to this group, which will be treated using radiofrequency (RF) ablation technique.
  Interventions: Device: Radiofrequency (RF)
- Cryotherapy (CRYO) (Active Comparator): Twenty patients will be allocated to this group, which will be treated using Cryotherapy (CRYO) ablation technique.
  Interventions: Device: Cryotherapy (CRYO)

INTERVENTIONS:
Device: Radiofrequency (RF) — Will be evaluated if percutaneous radiofrequency catheter ablation is superior to cryotherapy as treatment modality of para-hisian accessory pathways.
  Arms: Radiofrequency (RF)
Device: Cryotherapy (CRYO) — Will be evaluated if percutaneous cryotherapy catheter ablation is superior to radiofrequency as treatment modality of para-hisian accessory pathways.
  Arms: Cryotherapy (CRYO)

SUMMARY:
A randomized pilot study to evaluate safety and efficacy endpoints for treatment of para-hisian accessory pathways according to two different strategies of lesion formation.

These patients will be divided into 2 groups with different strategies of treatment: group 1 treated with radiofrequency (RF) ablation, group 2 with cryotherapy (CRYO).

The primary outcome will be the recurrence rate of accessory pathway conduction after one year of follow-up. Secondary endpoints will be immediate success and rate of permanent atrioventricular (AV) block.

DETAILED DESCRIPTION:
This is a randomized study on the safety and efficacy for percutaneous ablation of para-hisian accessory pathways according to two different modalities: radiofrequency (RF) or cryotherapy.

Thirty patients with symptomatic or high-risk para-hisian accessory pathways, documented by previous electrophysiological study (EPS), referred to percutaneous catheter ablation, will be enrolled in this trial.

After informed consent, these patients will be randomized in 2 groups with different current established strategies of invasive treatment. Group I: electrophysiological mapping and ablation with radiofrequency (RF) focal lesion formation.

Group II: electrophysiological mapping and ablation with cryotherapy (CRYO) focal lesion formation.

The primary outcome will be the recurrence rate of accessory pathway conduction after one year of follow-up. Secondary endpoints will be immediate success and rate of permanent atrioventricular (AV) block.

ELIGIBILITY:
Inclusion Criteria:

* Patients with para-hisian accessory pathways, diagnosed by electrophysiological study (EPS), with indication of invasive treatment according to current guidelines. Patients should be willing and able to sign an informed consent form, and to undergo all procedures described in both the study protocol and the consent form.

Exclusion Criteria:

* Previous cryotherapy ablation;
* Previous extensive radiofrequency ablation (including aortic cusp mapping);
* Age below twelve years;
* Severe coagulation disorder;
* Pregnancy;
* Refusal to participate in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
One-year recurrence rate | One year
  Recurrence rate of accessory pathway conduction, as assessed by follow-up Clinical recording and event monitoring external device (Holter/Looper).

SECONDARY OUTCOMES:
Immediate success rate | Time span between vein puncture (start of procedure) and sheath removal (end of procedure), comparing with baseline rhythm
  Mensuration of immediate success at the EP lab after ablation therapy is finished, defined by elimination of accessory pathway and/or noninducibility of arrhythmias at the end of procedure, as assessed by standard electrophysiological maneuvers.
  If an evidence of accessory pathway conduction still remains at the end of procedure it will count as an unsuccessful case.
  Does not take into account recurrences after the end of procedure, e.g. in the hospital ward before discharge.
Rate of atrioventricular block | up to 24 hours
  Safety outcome of any permanent atrioventricular (AV) block that occurred immediately after ablation start or during hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio I Scanavacca, MD, PhD, Study Chair — Instituto do coração - HC/FMUSP
Locations (1):
- Arrhythmia Clinical Unit - Instituto do Coração - HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No